CLINICAL TRIAL: NCT05968781
Title: A Prospective Observational Study of Predictive Factors for Successful Videolaryngoscopic Intubation Without Stylet
Brief Title: Predictive Factors for Successful Videolaryngoscopic Intubation Without Stylet
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: 2307-023-1443
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Intubation; Difficult or Failed; Videolaryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators aimed to evaluate the predictive factors for successful videolaryngoscopic intubation without stylet.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years and older
* Patients undergoing general anesthesia for elective surgery and requiring endotracheal intubation

Exclusion Criteria:

* Patients with suspected cervical spine injury
* Patients requiring rapid sequence induction and intubation.
* Patients with airway disorders
* Body Mass Index > 35 kg/m2
* Patients with a history of difficult intubation or, based on clinical judgment, anticipated difficult intubation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia and endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
First-pass success rate of videolaryngoscopic intubation without stylet | From the start of endotracheal intubation to 120 seconds
  An intubation attempt is defined as passing the laryngoscope blade between the patient's teeth. Duration of endotracheal intubation is defined from the moment the operator grasps the tube until the black line on the tube passes through the vocal cords

SECONDARY OUTCOMES:
Success rate of videolaryngoscopic intubation without stylet using BURP maneuver after failure of the first attempt | From the start of endotracheal intubation to 120 seconds
  An intubation attempt is defined as passing the laryngoscope blade between the patient's teeth. Duration of endotracheal intubation is defined from the moment the operator grasps the tube until the black line on the tube passes through the vocal cords
Incidence of using a stylet for the success of videolaryngoscopic intubation after the failure of the second attempt using the BURP maneuver | From the start of endotracheal intubation to 120 seconds
  An intubation attempt is defined as passing the laryngoscope blade between the patient's teeth. Duration of endotracheal intubation is defined from the moment the operator grasps the tube until the black line on the tube passes through the vocal cords
Incidence of successful endotracheal intubation after the failure of the third attempt using stylet | From the start of endotracheal intubation to 120 seconds
  An intubation attempt is defined as passing the laryngoscope blade between the patient's teeth. Duration of endotracheal intubation is defined from the moment the operator grasps the tube until the black line on the tube passes through the vocal cords
Time to completion of endotracheal intubation | From the start of endotracheal intubation to 120 seconds
  An intubation attempt is defined as passing the laryngoscope blade between the patient's teeth. Duration of endotracheal intubation is defined from the moment the operator grasps the tube until the black line on the tube passes through the vocal cords

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea